CLINICAL TRIAL: NCT05583409
Title: Effect of SBRT Combined With Osimertinib Compared With Osimertinib Alone for Stage IV Non-small Cell Lung Cancer
Brief Title: SBRT Combined With Osimertinib Compared With Osimertinib for Stage IV NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Li Zhang (Other)
Collaborators: Hubei Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC-LC002
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: SBRT plus Osimertinib versus Osimertinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osimertinib plus SBRT (Experimental): SBRT with photon and dose is 40Gy/5F after three months after Osimertinib treatment
  Interventions: Radiation: SBRT+Osimertinib
- Osimertinib (Active Comparator): Osimertinib 80mg, po, Qd
  Interventions: Drug: Osimertinib 80 MG

INTERVENTIONS:
Radiation: SBRT+Osimertinib — Received SBRT after three months of Osimertinib treatment
  Arms: Osimertinib plus SBRT
Drug: Osimertinib 80 MG — Osimertinib 80mg, po, Qd
  Arms: Osimertinib

SUMMARY:
This is a Prospective, Multicenter, Randomized Controlled study to evaluate Stereotactic Body Radiation Therapy (SBRT) as a potential treatment for stage IV non-small cell lung cancer (NSCLC) that has a mutated epidermal growth factor receptor (EGFR) and has been receiving treatment with Osimertinib

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy proven metastatic NSCLC (Stage IV).
2. Patients receiving first-line Osimertinib for EGFR mutant-positive for 3 months and achieved stable disease or partial response.
3. Age 18 to 75 years old.
4. Patients must have measurable disease at baseline.
5. The amount of metastatic focus <5.
6. ECOG score 0-2 7 Adequate normal organ and marrow function for TKI treatment and radiotherapy.

8. Patients must has sensitizing EGFR mutation (e.g. exon 19 deletion or exon 21 L858R) 9. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who previously received radiotherapy to the primary site.
2. Patient can't tolerate radiotherapy or targeted therapy;
3. Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  the time from the beginning of Osimertinib treatment to disease progression or death

SECONDARY OUTCOMES:
OS | 3 years
  the time from the beginning of Osimertinib treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD,PhD, Principal Investigator — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, 430030, Hubei, P. R. China, Wuhan, Hubei, China